CLINICAL TRIAL: NCT07124871
Title: Platelet Rich Plasma - Derived Exosomes Therapy for Erectile Dysfunction: A Feasibility Clinical Trial
Brief Title: PRP Exosomes Therapy for Erectile Dysfunction
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute for the Study of Urological Diseases, Greece (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRP-DET:7/3/25
Record Dates: First submitted 2025-04-27; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Erectile Dysfunction Due to Arterial Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental): All patients will be regular PDE5I users/responders. After one one-month washout period, ED patients will be screened by the IIEF-EF domain, and 30 eligible patients will be enrolled. subjects will receive three sessions of PRP-derived exosomes injection with 21± 3 days treatment interval.
  Interventions: Biological: PRP-derived exosomes injection

INTERVENTIONS:
Biological: PRP-derived exosomes injection — All subjects will receive three sessions of PRP-derived exosomes injection with 21± 3 days treatment interval.The patient will be positioned supine.
  A ¼-inch Penrose drain will be used as a tourniquet by placing it at the base of the penis and maintaining it in place under tension by a sterile clamp. We will obtain 10 mL of PRP per patient, but one of them will be used for platelet cell count analysis. A total 9 mL of the PRP-derived exosomes will be infused steadily over a 2 minutes period - 4.5 mL each into the right and left corpus cavernosum. The infusion will be performed at this slow speed - each side over 2 minutes of infusion - to minimize injury to the exosomes and cells. Following administration, compression of the penis will be achieved with a clenched fist for 20 minutes. At 20 minutes, the tourniquet will be removed, and a compressive dressing will be placed around the penile shaft. The patient will be instructed to remove the compression bandage in 4 hours

SUMMARY:
It will be a Single-arm, single-center, feasibility clinical trial with Primary Objective to investigate the treatment efficacy of PRP-derived exosomes injection in men with mild-moderate vasculogenic ED, as measured by the International Index of Erectile Function (IIEF). Also secondary objectives will be to study the adverse events and safety of the PRP-derived exosomes injection treatment in vasculogenic ED patients Study Centers The study will be carried out at Saint Lucas Hospital, Thessaloniki, Greece. Laboratory tests of all patients will be performed at the hospital's microbiology laboratory. PRP-derived exosomes preparation and application will take place at the Regenerative Clinic.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate.
* Age 40-70 years.
* Sexually active in a stable, heterosexual relationship of more than three months duration.
* Presence of ED for at least 6 months.
* IIEF-ED: 17-25 at visit 2. The IIEF classifies the severity of ED into five categories stratified by score: No ED: 26-30, Mild ED: 22-25, Mild to moderate ED: 17-21, Moderate ED: 11-16 and Severe ED: 6-10.
* Patients will be PDE5i users for at least 6 months and report some/good response to PDE5i in the last month before screening (at visit 1
* Agree to suspend all ED therapy for the duration of the study.
* Agree to attempt sexual intercourse at least 4 times every 3 weeks for the duration of the study without being under the influence of alcohol or recreational drugs.
* Agree to document the outcome using IIEF questionnaire during every visit and the Sexual Encounter Profile (SEP) diary, as needed (months 1 and 3 post treatment).

Exclusion Criteria:

* Previous major pelvic surgery or pelvic trauma that could impact EF, such as radical prostatectomy, radical cystectomy, or rectal surgery. 19
* Patients with previous transurethral resection of the prostate (TURP) surgery without sequelae of iatrogenic ED may be included.
* Previous penile surgery of any kind except circumcision and condyloma removal, such as penile lengthening, penile cancer surgery, penile plication, and grafting.
* Previous history of priapism or penile fracture
* Previous radiation therapy to the pelvis.
* Abnormal morning serum testosterone level, defined as a value lower than 300 ng/dL (indicative of untreated hypogonadism) or greater than1197 ng/dL.
* Current or previous hormone use, other than prescribed testosterone, clomiphene or thyroid medication. Subjects with prior or current use of hormonal treatment for prostate cancer are also excluded.
* Psychogenic ED.
* Peyronie's Disease or penile curvature that negatively influences sexual activity.
* Anatomical or neurological abnormalities in the treatment area.
* Any untreated medical condition (based on medical history)
* Patients with generalized polyneuropathy or neurological conditions irrespective of cause, such as severe diabetes, multiple sclerosis, or Parkinson's Disease.
* Refusal to suspend ED therapy for the duration of the study. Subjects who are using Tadalafil as a treatment for benign prostatic hyperplasia (BPH) will also be excluded.
* Men deemed not healthy enough to participate in sexual activity.
* Any condition or behavior that indicates to the Principal Investigator that the subject is unlikely to be compliant with study procedures and visits.
* Any health history or laboratory result that indicates to the Principal Investigator that the subject has a significant medical condition and should not participate in the study.
* History of consistent treatment failure with PDE5 inhibitors for therapy of ED.
* Any history of significant psychiatric diseases, such as bipolar disorder or psychosis, greater than one lifetime episode of major depression, current depression of moderate or greater severity.
* Patients who are currently using SSRI or psychotropic medications.
* Partners who are < 18 years of age, who are nursing, who wish to become pregnant during the study period, and who have any gynecologic problems, sexual dysfunction, or major medical conditions that would limit participation in sexual intercourse.
* Patients with any hematological disorder

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The % of patients in each group who attain Minimal Clinically Important Difference (MCID) in the International Index for Erectile Function- Erectile Function (IIEF-EF) domain | From baseline to 12 weeks after final treatment
  The IIEF classifies the severity of ED into five categories stratified by score: No ED: 26-30, Mild ED: 22-25, Mild to moderate ED: 17-21, Moderate ED: 11-16 and Severe ED: 6-10.
  MCID values for the IIEF-EF (Erectile Function) domain are 2-point increase for mild ED, a 5-point increase for moderate ED and a 7-point increase for severe ED In IIEF-EF score higher values mean better outcome

SECONDARY OUTCOMES:
The % of patients who attain Minimal Clinically Important Difference(MCID) in the International Index for Erectile Function- Erectile Function (IIEF-EF) domain . | From baseline to 4 weeks after final treatment
  The IIEF classifies the severity of ED into five categories stratified by score: No ED: 26-30, Mild ED: 22-25, Mild to moderate ED: 17-21, Moderate ED: 11-16 and Severe ED: 6-10.
  MCID values for the IIEF-EF (Erectile Function) domain are 2-point increase for mild ED, a 5-point increase for moderate ED and a 7-point increase for severe ED In IIEF-EF score higher values mean better outcome
The change of the International Index for Erectile Function- Erectile Function (IIEF-EF) domain from baseline to 12 weeks after final treatment. | From baseline to 12 weeks after final treatment.
  The IIEF classifies the severity of ED into five categories stratified by score: No ED: 26-30, Mild ED: 22-25, Mild to moderate ED: 17-21, Moderate ED: 11-16 and Severe ED: 6-10.
  MCID values for the IIEF-EF (Erectile Function) domain are 2-point increase for mild ED, a 5-point increase for moderate ED and a 7-point increase for severe ED In IIEF-EF score higher values mean better outcome
Adverse events in all patients | Periprocedural

CONTACTS AND LOCATIONS:
Locations (1):
- St Lukes Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colombo M, Raposo G, Thery C. Biogenesis, secretion, and intercellular interactions of exosomes and other extracellular vesicles. Annu Rev Cell Dev Biol. 2014;30:255-89. doi: 10.1146/annurev-cellbio-101512-122326. Epub 2014 Aug 21. PMID 25288114